CLINICAL TRIAL: NCT01231451
Title: The Pharmacokinetics of Depot Medroxyprogesterone Acetate (DMPA) in the Absence and Presence of Lopinavir/Ritonavir in HIV-1 Infected Women
Brief Title: Depot Contraception With and Without Lopinavir/Ritonavir
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Ethics board said the study could not be fully justified.
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Laura Waters, St Stephen's AIDS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SSAT 038
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infection
Keywords: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — N,N-dimethyl-4-anisidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): All Subjects will receive the same intervention
  Interventions: Drug: DMPA

INTERVENTIONS:
Drug: DMPA — All subjects will take DMPA

SUMMARY:
DMPA (depot medroxyprogesterone acetate or the 'depot' injection) is a widely used contraception. It is popular in woman with HIV as it probably still works when you take HIV drugs. HIV drugs can increase or decrease the level of other drugs (e.g. contraceptives) in your bloodstream which may make them work less well or increase side effects. It is assumed that DMPA can be given with HIV drugs there are no studies proving this.

The purpose of the study is to investigate whether an HIV drug combination containing lopinavir/ritonavir affects DMPA when they are taken at the same time.

DETAILED DESCRIPTION:
Lopinavir/ritonavir (LPV/r) is licensed for use in combination with other antiretrovirals for the treatment of HIV infection. Like other agents from the protease inhibitor class, LPV/r inhibits the 3A isoenzyme of the hepatic cytochrome P450 system and may increase the levels of drugs metabolised via this route. However, LPV/r has also been shown in vivo to induce its own metabolism and to increase the biotransformation of some drugs metabolized by P450 enzymes and by glucuronidation.

Women account for an increasing proportion of the HIV epidemic in the UK. The huge reductions in HIV-related mortality and morbidity associated with the use of effective combination antiretroviral therapy have led to a shift in focus to longer term issues, including reproductive health and contraception. The impact of a variety of antiretrovirals on the plasma pharmacokinetics of oral oestrogen and progesterone preparations have been investigated and in general NNRTIs and boosted PIs cause a reduction in levels of both, particularly oral oestrogen preparations. Most package inserts for combined (oestrogen and progestogen) and progestogen-only oral contraceptives recommend that additional contraceptive methods be employed with concomitant use of enzyme-inducing agents.

Injectable contraception provides highly effective contraception without the need for daily pill taking, an important factor to consider for individuals already taking regular medication. Depot medroxyprogesterone acetate (DMPA) is the most frequently prescribed injectable method. DMPA, like other progestogens, is metabolised by the cytochrome P450 system but interaction studies in women on antiretrovirals are limited. A study of 59 women on DMPA contraception plus an unboosted PI (nelfinavir) or an NNRTI (efavirenz or nevirapine) measured DMPA levels and compared them with 16 women on either no therapy or NRTIs only (no potential for drug interaction). DMPA levels were similar in all groups and suppression of ovulation over a 12 week period was also similar in all groups.

Although the high levels of DMPA achieved over the dosing interval make any pharmacokinetic interaction unlikely to be clinically significant, some clinicians advise a reduction in the interval between DMPA injections from 12 to 10 weeks in patients on an NNRTI or boosted PI; there is no clear evidence to support this approach. Although the described study supports normal dosing intervals for women on an NNRTI, the unboosted PI nelfinavir is not recommended as standard of care and the impact of ritonavir-boosted PIs is unclear. The summary of product characteristics for DMPA advises a normal dosing interval even when using a potent enzyme inducers, suggesting no additional intervention is required when prescribing a boosted PI. Formal pharmacokinetic data is crucial to clarify this important area.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
2. Non-pregnant, non-lactating premenopausal females.
3. No current hormonal contraception (short acting methods eg oral contraceptive pills and patches can be removed at screening)
4. Regular menstrual periods such that DMPA can be administered between days 1-5 of menstrual cycle
5. Between 18 and 45 years, inclusive.
6. Documented HIV-1 infection
7. Must be willing to use a barrier method of contraception to avoid pregnancy throughout the study, and for at least 56 days following completion of the study.
8. CD4 count > 200 at screening (Note: retesting of screening CD4 count allowed).
9. Clinician and patient happy to delay HAART until week 12 of study
10. Not currently on HAART and eligible to receive LPV/r and Truvada as determined by their primary HIV care provider in accordance with treatment guidelines
11. If history of HAART exposure, no virological failure (prior drug switches allowed if for tolerability/toxicity/convenience of dosing).
12. Agrees not to change regimen, outside the study recommendations, from baseline until end of the treatment period unless this is medically indicated as decided by the treating physician

Exclusion Criteria:

1. Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance with the protocol. This would include any active clinically significant renal, cardiac, hepatic, pulmonary, vascular, metabolic disorders or malignancy.
2. Have a body mass index (BMI) >35
3. Personal history of venous thromboembolism (VTE) or pulmonary embolism (PE)
4. Presence of any current active AIDS defining illness (Category C conditions in the CDC Classification System for HIV 1993) except stable cutaneous Kaposi's Sarcoma
5. Osteoporosis or significant risk factors for osteoporosis (alcohol abuse, long-term anticonvulsants/corticosteroids, BMI less than 18, eating disorder, previous low trauma fracture, significant family history osteoporosis)
6. Conditions for which DMPA is contra-indicated or risks outweigh benefits:

   1. Significant multiple risk factors for arterial cardiovascular disease
   2. Vascular disease
   3. Previous or current venous thromboembolism (VTE) or pulmonary embolism (PE)
   4. Ischaemic heart disease
   5. Stroke (history of cerebrovascular accident)
   6. Headaches migraine with aura, at any age
   7. Unexplained vaginal bleeding
   8. Gestational trophoblastic neoplasia (GTN) (includes hydatidiform mole, invasive mole, placental site trophoblastic tumour) hCG abnormal
   9. Breast cancer (past or current) or strong family history
   10. Diabetes nephropathy/retinopathy/neuropathy
   11. Other vascular disease or diabetes of >20 years' duration
   12. Viral hepatitis (active)
   13. Presence or history of any sever hepatic disease where liver function tests have not returned to normal
   14. Cirrhosis (decompensated)
7. Clinically relevant alcohol or drug use (positive urine drug screen, excluding cannabinoids) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
8. The use of disallowed concomitant therapy (See section 5.2).
9. Previous allergy to any of the constituents of the study pharmaceuticals.
10. Exposure to any investigational drug or placebo within 4 weeks of baseline.
11. Any HAART exposure within 6 months of screening for this study (ie participants need to be treatment-naïve or on a treatment interruption for 6 months or more).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetics of depot medroxyprogesterone acetate (DMPA) | week 1 - week 24
  To investigate the pharmacokinetics of depot medroxyprogesterone acetate (DMPA) in the absence and presence of lopinavir/ritonavir in HIV-
  1 infected women

SECONDARY OUTCOMES:
Impact of co-administration of DMPA and lopinavir/ritonavir | Week 1 - week 24
  To investigate the impact of co-administration of DMPA and lopinavir/ritonavir on surrogate markers of contraceptive efficacy (LH, FSH, oestradiol)
Safety of DMPA | Week 1 - week 24
  To investigate the safety of DMPA in HIV infected women on lopinavir/ritonavir
Impact of DMPA on lopinavir/ritonavir plasma concentrations | week 1 - week 24
  To investigate the impact of DMPA on lopinavir/ritonavir plasma concentrations compared with historical controls

CONTACTS AND LOCATIONS:
Locations (1):
- St Stephen's Centre, London, United Kingdom